CLINICAL TRIAL: NCT05313035
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Immunogenicity of SARS-CoV-2 Protein Subunit Recombinant Vaccine (Bio Farma) Adjuvanted With Alum+CpG 1018 in Healthy Populations Aged 18 Years and Above in Indonesia
Brief Title: Safety and Immunogenicity Study of COVID-19 Protein Subunit Recombinant Vaccine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Indonesia University (Other); Faculty of Medicine, Diponegoro University, Semarang (Unknown); Faculty of Medicine, Universitas Andalas, Padang (Unknown); Faculty of Medicine, Universitas Hassanudin, Makassar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CoV2-020322
Record Dates: First submitted 2022-04-05; First posted 2022-04-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; healthy population
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Vaccine candidate and placebo are masking, lot number is masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vaccine Candidate Formula 1 (Experimental): 2 doses of vaccine candidate formula 1 administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 protein subunit recombinant vaccine
- Vaccine Candidate Formula 2 (Experimental): 2 doses of vaccine candidate formula 2 administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 protein subunit recombinant vaccine
- Control (Placebo Comparator): 2 doses of placebo administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: SARS-CoV-2 protein subunit recombinant vaccine — candidate vaccine manufactured by PT. Bio Farma
  Arms: Vaccine Candidate Formula 1; Vaccine Candidate Formula 2
Biological: placebo — the placebo is NaCl injection manufactured by PT. Bio Farma
  Arms: Control

SUMMARY:
This trial is observer-blind, comparative, randomized, placebo-controlled phase 2 study. The population is healthy subjects aged 18 and above

DETAILED DESCRIPTION:
The phase 2 is dose-ranging study which will recruit 360 subjects to compare two vaccine formulas to placebo (1:1:1), to evaluate the safety and immunogenicity of the vaccine. The subjects will be given 2 doses of investigational product with 28 days interval between doses.

One selected vaccine formula will be evaluated for safety and persistence antibody until 6 months after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy subjects aged 18 years and above.
2. Subjects have been informed properly regarding the study and signed the informed consent form.
3. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. History of vaccination with any COVID-19 vaccine.
3. History of COVID-19 within 1 month (for mild-moderate disease) or 3 months (for severe disease) prior to enrollment.
4. Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
5. Women who are pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).
6. History of uncontrolled asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
7. History of blood disorders contraindicating intramuscular injection.
8. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc) which according to the investigator might interfere with the assessment of the trial objectives.
9. History of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immuneresponse (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
10. History of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre syndrome.
11. Subjects receive any vaccination (other than COVID-19 vaccine) within 1 month before and after IP immunization.
12. Subjects plan to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of the candidate vaccine | 14 days after the last dose
  seroconversion rate of antibody (IgG and neutralization antibody)

SECONDARY OUTCOMES:
Safety of the candidate vaccine | 28 days after each dose
  percentage of subjects with solicited and unsolicited Adverse Events (AE)
Serious Adverse Event (SAE) of the vaccine | 6 months after the last dose
  percentage of subjects with at least 1 SAE
Persistence antibody of vaccine candidate | 14 days, 28 days, 3 months, 6 months after the last dose
  GMT of antibody (IgG and neutralization antibody)
Persistence antibody of vaccine candidate | 14 days, 28 days, 3 months, 6 months after the last dose
  seropositive rate of antibody (IgG and neutralization antibody)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Soedjatmiko SpA(K), MSi, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (3):
- Indonesia (3):
  - Faculty of Medicine, Diponegoro University, Semarang, Semarang, Central Java
  - Faculty of Medicine Universitas Hassanudin, Makassar, South Sulawesi
  - Faculty of Medicine, Universitas Andalas, Padang, Padang, West Sumatera